CLINICAL TRIAL: NCT01468701
Title: GLORIA - AF: Global Registry on Long-Term Oral Anti-thrombotic Treatment In Patients With Atrial Fibrillation (Phase II/III)
Brief Title: GLORIA-AF Registry Program - Second and Third Phases
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.129
Record Dates: First submitted 2011-10-28; First posted 2011-11-09 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this part of the Registry Program patients with non-valvular atrial fibrillation (AF) at risk for stroke are enrolled to characterize the target population and to collect real world data on important outcome events. For administrative purposes the study is divided into two protocol numbers: 1160.129 for all non-EU (European Union) and non-EEA (European Economic Area) countries, and 1160.136 for EU and EEA countries. The total number of patients enrolled in both protocols is estimated to be 48,000 patients, and all these patients will be included in the data analysis for study 1160.129.

ELIGIBILITY:
Inclusion criteria:

1. Age =>18 years at enrollment
2. Male or female patient (or legally acceptable representative) willing and able to provide written informed consent
3. Patient newly diagnosed (< 3 months prior to baseline visit) with non-valvular AF and at risk for stroke.

Other inclusion criteria apply.

Exclusion criteria:

1. Presence of any mechanical heart valve, or valve disease that is expected to require valve replacement intervention;
2. Patients who have received more than 60 days of vitamin K antagonist (VKA) treatment in their lifetime;
3. AF with a generally reversible cause;
4. Patients with a medical condition other than atrial fibrillation for which chronic use of an oral anticoagulant (for example, a VKA) is indicated Other exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-valvular AF
Sampling Method: Non-Probability Sample
Enrollment: 37235 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (665):
- United States (323):
  - University South Alabama Medical Center, Mobile, Alabama
  - Black Warrior Research, Northport, Alabama
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Phoenix Heart PLLC, Glendale, Arizona
  - Mercy Cinic Hot Springs Communities, Hot Springs, Arizona
  - Midwest Internal Medicine, PLLC, Lake Havasu City, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Dr. Michael A. Frais, Cardiologist, P.A., Hot Springs, Arkansas
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Donald W. Reynolds Institute on Aging, Little Rock, Arkansas
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Diagnamics, Inc, Encinitas, California
  - Allianz Medical and Research Center, Fountain Valley, California
  - B&K Medical Research Center, Fresno, California
  - American Clinical Trials, Hawaiian Gardens, California
  - Scripps Clinic, La Jolla, California
  - La Mesa Cardiac Center, La Mesa, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Mehrdad Kevin Ariani, MD, Incorporated, Northridge, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - Ritchken and First MD's, San Diego, California
  - Coastal Heart Group Inc, Santa Ana, California
  - Pacific Heart and Vascular, Stockton, California
  - Southwest Heart Institute, Temecula, California
  - University of California Los Angeles, Torrance, California
  - Cardiology Associates Medical Group Inc, Ventura, California
  - Ventura Cardiology Consultants Medical Group, Inc, Ventura, California
  - Ventura Clinical Trials, Ventura, California
  - Office of Dr. David J Cislowski MD, Visalia, California
  - Aurora Denver Cardiology Associates, PC, Aurora, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Connecticut Heart and Vascular Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Associates of Fairfield County, Norwalk, Connecticut
  - Norwalk Medical Group, Norwalk, Connecticut
  - Heart Specialists, PC of Southern CT, Shelton, Connecticut
  - Red Clay Research LLC., Newark, Delaware
  - Howard University Hospital, Washington D.C., District of Columbia
  - Cardiac Arrhythmia Center, Washington D.C., District of Columbia
  - Medical Faculty Associates, Inc, Washington D.C., District of Columbia
  - Aventura Institute for Cardiovascular Wellness, PA, Aventura, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Seidman Clinical Trials, Delray Beach, Florida
  - Universal Clinical Research Associates, Doral, Florida
  - Cardiovascular Research of North Florida LLC, Gainesville, Florida
  - Magi Research Clinic, Inc, Hialeah, Florida
  - Global Research Solutions Corporation, Hollywood, Florida
  - St. Vincent's Ambulatory Care, Jacksonville, Florida
  - Tenet Florida Physician Services, Jupiter, Florida
  - Watson Clinic Center for Research, Inc, Lakeland, Florida
  - A&L Clinical Research, Miami, Florida
  - Miami Center for Cardiovascular Disease, Miami, Florida
  - Global Research Solutions Corporation, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Sacred Heart Medical Specialty Group, Miramar Beach, Florida
  - Collier HMA Physician Management, Naples, Florida
  - Edgewater Medical Research, New Smyrna Beach, Florida
  - SouthEast Medical Centre, Oakland Park, Florida
  - Research One, Orlando, Florida
  - South Florida Research Solutions, LLC, Pembroke Pines, Florida
  - Langhorne Cardiology Consultants, Inc, Pensacola, Florida
  - VNH Heart Center Research, Port Charlotte, Florida
  - Brevard Cardiovascular Research Associates, Inc, Rockledge, Florida
  - Velella Research, Inc, Sarasota, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - James C. Neiman, MD, Seminole, Florida
  - Suncoast Cardiovascular Research Inc., St. Petersburg, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Alternative Solutions Medical Research and Prevention Center, St. Petersburg, Florida
  - Tallahassee Research Instutite, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Indian River Medical Associates Cardiology, Vero Beach, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Executive Health and Research Associates, Atlanta, Georgia
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - Atlanta Heart Specialists, LLC, Cumming, Georgia
  - William C McGarity, Jr, MD, PC, Decatur, Georgia
  - Coliseum Medical Center, Macon, Georgia
  - Kootenai Heart Clinics, LLC, Coeur d'Alene, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Prairie Cardiovascular Memorial Hospital, Carbondale, Illinois
  - Captain James A. Lovell Federal Health Care Center, Chicago, Illinois
  - Medex Healthcare Research, Chicago, Illinois
  - John H. Stroger Jr. Hospital of Cook Country, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - North Shore Cardiology Consultants, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Advanced Heart Care, LLC, Medicoricum, LLC, Fairview Heights, Illinois
  - Adventist Health Partners, Inc, Hinsdale, Illinois
  - Consultants in Cardiovascular Medicine, Melrose Park, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Advanced Cardiovascular Consultants, Rock Island, Illinois
  - DuPage Medical Group, Winfield, Illinois
  - Hendricks Family Medicine, Brownsburg, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Beacon Medical Group Clinical Research, La Porte, Indiana
  - Cardiology Associates of Northwest Indiana, PC, Munster, Indiana
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Central Cardiology Associates, Elizabethtown, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Baptist Health Clinical Studies, Madisonville, Kentucky
  - Office of Dr. Paul McLaughlin, M.D., Mount Sterling, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Grace Research, LLC, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Cardiovascular Specialists of Southwest Louisiana, LLC, Lake Charles, Louisiana
  - Medpharmics, LLC, Metairie, Louisiana
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Southern Maine Health Care, Biddeford, Maine
  - Cardiac Consultants, LLC, Annapolis, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Cardiovascular Specialists of Central Maryland, Columbia, Maryland
  - Delmarva Heart Research Foundation, Inc, Salisbury, Maryland
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - Chesapeake Cardiovascular Associates, Towson, Maryland
  - Primary Care Cardiology Research, Inc, Ayer, Massachusetts
  - Genesys Research Institute, Incorporated, Brighton, Massachusetts
  - NECCR Internal Med and Cardio, Fall River, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Endeavor Medical Research, Alpena, Michigan
  - McLaren Bay Region Medical Center, Bay City, Michigan
  - Henry Ford Hospital K-15, Detroit, Michigan
  - St. Vincent Consultants in Cardiovascular Disease, LLC, Erie, Michigan
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Genesys Heart Institute, Grand Blanc, Michigan
  - Regional Cardiology Associates, Grand Blanc, Michigan
  - Thoracic and Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Upper Michigan Cardiovascular Associates, PC, Marquette, Michigan
  - McLaren-Macomb, Mount Clemens, Michigan
  - South Western Medical Clinic, Niles, Michigan
  - Providence Park Hospital, Novi, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - MId-MIchigan Heart and Vascular Center, Saginaw, Michigan
  - Essentia Heart and Vascular Clinic, Duluth, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - The Center for Clinical Trials, Inc., Biloxi, Mississippi
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Health Midwest Ventures Group, Inc, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Louis University, St Louis, Missouri
  - Consult and Research Associates, St Louis, Missouri
  - Gateway Cardiology, PC, St Louis, Missouri
  - Kalispell Regional Medical Center, Kalispell, Montana
  - MidAmerica Cardiovascular Institute, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Board of Regents of the University of Nebraska, Omaha, Nebraska
  - Alegent Health Heart and Vascular Specialists, Papillion, Nebraska
  - Renown Institute for Heart and Vascular Health, Reno, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Medicor Cardiology, Bridgewater, New Jersey
  - Cooper University Hospital, Camden, New Jersey
  - Monmouth Cardiology Associates, Eatontown, New Jersey
  - Electrophysiology Associates of Northern New Jersey, Hackensack, New Jersey
  - Advocare Heights Primary Care, Haddon Heights, New Jersey
  - Associated Cardiovascular Consultants Lourdes, Hammonton, New Jersey
  - NJ Heart LLC, Linden, New Jersey
  - Garden State Heart Care, PC, Manalapan, New Jersey
  - Atlantic Cardiology, LLC, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Heart and Vascular Center of New Brunswick, Somerset, New Jersey
  - Central New Jersey Cardiology, South Plainfield, New Jersey
  - Associated Cardiovascular Consultants Lourdes, Voorhees Township, New Jersey
  - NJ Cardiology Associates, West Orange, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Albany Medical Center / Albany Medical College, Albany, New York
  - New York -Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Community Cardiology, Camillus, New York
  - Bassett Medical Center, Cooperstown, New York
  - New York Hospital Queens, Flushing, New York
  - UHS Office of Clinical Trials, Johnson City, New York
  - Long Island Heart Associates, Mineola, New York
  - Chinatown Cardiology, PC, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Saint Luke - Roosevelt Hospital Center, New York, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Stony Brook Cardiology/Electrophysiology, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Heart Center, Syracuse, New York
  - Cardiac Care and Vascular Medicine, PLLC, The Bronx, New York
  - Great Lakes Medical Research, Westfield, New York
  - Cardiology Group of Western New York, PC, Williamsville, New York
  - Kernodle Clinic West, Burlington, North Carolina
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - Carolina Cardiology Cornerstone, High Point, North Carolina
  - Profen Research Network at East Carolina Medical Associates, Jacksonville, North Carolina
  - Kannapolis Internal Medicine, Kannapolis, North Carolina
  - Clinical Trials of America, Inc, Lenoir, North Carolina
  - Pinehurst Medical Clinic, Inc, Pinehurst, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Wake Heart and Vascular Associates, Wilson, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Trinity Health Center Medical Arts, Minot, North Dakota
  - Aultman Hospital, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Mercy Health Fairfield Hospital, Fairfield, Ohio
  - Cleveland Cardiovascular Research Foundation, Fairview Park, Ohio
  - Emil Hayek, M.D., Inc, Hudson, Ohio
  - Innovation Center, Kettering Medical Center, Kettering, Ohio
  - RAS Health Ltd, Marion, Ohio
  - Frederick C Smith Clinic Inc, Marion, Ohio
  - Mound Family Practice, Miamisburg, Ohio
  - Heart House Research Foundation, LLC, Springfield, Ohio
  - Cardiovascular Research Center, Toledo, Ohio
  - Toledo Clinic Incorporated, Toledo, Ohio
  - Great Lakes Medical Research, LLC, Willoughby, Ohio
  - Ohio Heart Institute, Youngstown, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - INTEGRIS Ambulatory Care Corporation, Yukon, Oklahoma
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - Fanno Creek Clinic, LLC, Portland, Oregon
  - Sacred Heart Medical Center at RiverBend, Springfield, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Preferred Primary Care Phys, Carnegie, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Physician Specialist of Northern Lancaster County Medcl Grp, Ephrata, Pennsylvania
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Lycoming Internal Medicine, Inc, Jersey Shore, Pennsylvania
  - Cardiology Consultants of Philadelphia, Lansdale, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Cardiology Associates, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Neurology Associates, Pittsburgh, Pennsylvania
  - Grand View - Lehigh Valley Health Services, Sellersville, Pennsylvania
  - Warminster Medical Associates, PC, Warminster, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - South County Cardiology, Wakefield, Rhode Island
  - AnMed Health Clinical Research, Anderson, South Carolina
  - Internal Medicine Associates of Anderson, PA, Anderson, South Carolina
  - Lowcountry Medical Group, LLC, Beaufort, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Piedmont Cardiology Associates, P.A., Greenwood, South Carolina
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Office of Yvonne Chester, Chattanooga, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Center For Cardiovascular Research, Johnson City, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - THV Research, LLC, Austin, Texas
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Heartplace, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Amir Malik Research, Fort Worth, Texas
  - State of the Heart Cardiology, Grapevine, Texas
  - Angiocardiac Care of Texas, Houston, Texas
  - Houston Methodist DeBakey Cardiology Associates, Houston, Texas
  - Barry Troyan, M.D, PA, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Dairy Ashford Family Pratice, Houston, Texas
  - Cardiovascular Associates PLLC, Humble, Texas
  - Cardiology Center of Houston, PA, Katy, Texas
  - Texas Cardiology Research Center PLLC, Kingwood, Texas
  - Caprock Cardiac Center Research Institute, Lubbock, Texas
  - Mission Research Institute, LLC, New Braunfels, Texas
  - Mercury Medical ,LLC, San Antonio, Texas
  - Texas Medical Research Associates, San Antonio, Texas
  - Sealy Urgent Care Center and Medical Clinic, Sealy, Texas
  - Seguin Institute of Cardiovascular Research, Seguin, Texas
  - Sugarland Cardiology, Sugar Land, Texas
  - Cardiovascular Associates of East Texas, PA, Tyler, Texas
  - Trinity Clinic, Tyler, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Providence Health Services of Waco, Waco, Texas
  - Hill County Primary Care, Whitney, Texas
  - Heart Center at Saint Mark's, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Cardiovascular Associates, Ltd, Chesapeake, Virginia
  - Cardiology Consultants of Danville, Inc, Danville, Virginia
  - Inova Research Center, Falls Church, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Mary Washington Hospital Research Department, Fredericksburg, Virginia
  - Harrisonburg Medical Associates, Harrisonburg, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Cardiovascular Associates of Virginia, Midlothian, Virginia
  - CJW Medical Center - Chippenham, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Selma Medical Associates, Winchester, Winchester, Virginia
  - Sound Medical Research, Port Orchard, Washington
  - The Polyclinic, Seattle, Washington
  - Franciscan Heart and Vascular Associates, Tacoma, Washington
  - Cardiac and Thoracic Institute of Central Washington, Yakima, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - University Cardiovascular Services, Huntington, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Mayo Clinic-Sparta, La Crosse, Wisconsin
  - Karim Bakhtiar MD, SC, Milwaukee, Wisconsin
  - Family Medical Clinic, Milwaukee, Wisconsin
  - Wheaton Franciscan, Milwaukee, Wisconsin
  - Milwaukee VA Medical Center, Milwaukee, Wisconsin
  - ProHealth Care Research Institute and Cardiology Associates, Waukesha, Wisconsin
- Argentina (16):
  - Consultorios Hematologicos SRL, Buenos Aires
  - Clinica Coronel Suárez, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires
  - Instituto Cardiovascular de Corrientes Juana Francisca Cabra, Corrientes
  - Hospital Espanol de Mendonza, Godoy Cruz
  - Hospital Privado de Comunidad, Mar del Plata
  - DIM Clinica Privada, Ramos Mejía
  - Hospital Privado de Rosario, Rosario
  - Consultorio del Dr. Aiub, San Isidro
  - Sanatorio San Lucas, San Isidro
  - Sanatorio 9 de Julio S.A., San Miguel de Tucumán
  - Centro Privado de Cardiología, San Miguel de Tucumán
  - Unidad Coronaria San Geronimo S.R.L., Santa Fe
  - Clinical Juncal, Temperley
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Brazil (30):
  - Hospital Vera Cruz, Belo Horizonte
  - Clinica Procardio Ltda, Blumenau
  - Hospital do Coracao do Brasil, Brasília
  - Instituto de Cardiologia do Distrito Federal, Brasília
  - Hospital Angelina Caron, Campina Grande do Sul
  - Centro Especializado em Cardiol Loema Instituto de Pesq Clin, Campinas
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas
  - Hospital Nossa Senhora de Pompeia, Caxias do Sul
  - Irmandade da Santa Casa de Misericordia de Curitiba, Curitiba
  - Barroso e Sebba Ltda, Goiânia
  - CLINICOR-Clinica de Exames Cardiolog e Ecografias S S LTDA, Maceió
  - Hospital São Vicente de Paulo, Passo Fundo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Fundacao Universitaria de Cardiologia - Inst de Cardiologia, Porto Alegre
  - Pronto Socorro Cardiológico de Pernambuco Prof. Luiz Tavares, Recife
  - Hospital Copa D'or, Rio de Janeiro
  - Fundacao Pro-Coracao FUNDACOR, Rio de Janeiro
  - Instituto Cardiopulmonar da Bahia LTDA, Salvador
  - Fundacao Bahiana de Cardiologia, Salvador
  - Instituto de Ensino E Pesquisa Do Hospital Da Bahia, Salvador
  - Instituto de Molestias Cardiovasculares - IMC, São José do Rio Preto
  - H.S.J. Beneficência Portuguesa - São Paulo, São Paulo
  - FGM - Clínica Paulista de Doenças Cardiovasculares, São Paulo
  - Hcor - Hospital do Coracao, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina - FMUSP, São Paulo
  - Hospital Santa Marcelina, São Paulo
  - Hospital Sao Paulo UNIFESP, São Paulo
  - Instituto de Molestias Cardiovasculares Tatui SP, Tatuí
  - Santa Casa de Votuporanga, Votuporanga
- Canada (37):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - North Road Clinical Research, Coquitlam, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - Crestwood Med & Dental Bldg, Richmond, British Columbia
  - Ocean West Research Clinic Inc., Surrey, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Q & T Research Chicoutimi Inc, Chicoutimi, Migration Data
  - CardioVasc HR Inc., St-Jean-sur-Richel, Migration Data
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Eastern Health (MUN), St. John's, Newfoundland and Labrador
  - Antigonish Medical Associates Inc., Antigonish, Nova Scotia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cambridge Cardiac Care Inc., Cambridge, Ontario
  - West Lincoln Memorial Hospital, Grimsby, Ontario
  - Winterberry Family Medicine, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Victoria Hospital (LHSC), London, Ontario
  - Mississauga Clinical Research Centre, Mississauga, Ontario
  - SKDS Research Incorporated, Newmarket, Ontario
  - M Heffernan Medicine Professional Corp., Oakville, Ontario
  - Oshawa Clinic Cardiology Department, Oshawa, Courtice, Oshawa, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - University of Ottawa Heart Institute Cardiology Research, Ottawa, Ontario
  - Aviva Clinical Trial Group Inc., Stoney Creek, Ontario
  - SGH Medical Mall, Toronto, Ontario
  - Keele Medical Place, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique de Cardiologie de Levis, Lévis, Quebec
  - CHUM Hotel Dieu, Montreal, Quebec
  - Recherche Clinique Sigma Inc., Québec, Quebec
  - IUCPQ (Laval University), Sainte-Foy, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
  - Baycole Research, Saskatoon, Saskatchewan
- Chile (6):
  - Hospital Clínico Fuerza Aérea de Chile, Santiago
  - Centro de Estudios Clinicos Barros Luco, Santiago
  - Hospital y CRS El Pino, Santiago
  - CECMI Ltda, Temuco
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
  - Clinica Tabancura, Vitacura
- China (59):
  - Beijing AnZhen Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Beijing Shijingshan Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - 2nd Xiangya Hospital of Central South University, Changsha
  - Chinese Traditional Medicine Hospital of Sichuna Provinc, Chengdu
  - Center Hospital of Dalian, Dalian
  - Foshan Hospital of Southern Medical University, Foshan
  - Fujian Provincal Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - Wu Jing Zong Dui Hospital of Guangdong Province, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Shandong Jiaotong Hospital, Jinan
  - Center Hospital of Jinan, Jinan
  - Qianfoshan Hospital affiliated to Shandong University, Jinan
  - Shandong Provincial Hospital, Jinan
  - Jining No.1 people's hospital, Jining
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - QingDao Municipal Hospital, Qingdao
  - Qingdao Fuwai Hospital, Qingdao
  - Qingdao Central Hospital, Qingdao
  - Chinese People's Liberation Army 401 Hospital, Qingdao
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai Huadong Hospital, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - Shanghai East Hospital, Tongji University China, Shanghai
  - Renji Hospital Shanghai Jiaotong Univesrity School of Medicine, Shanghai
  - Minhang District Central Hospital, Shanghai
  - Songjiang Hospital, Shanghai
  - Jiading Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - General Hospital of Shenyang Military Region, Shenyang
  - People's Hospital of Liaoning Province, Shenyang
  - The Forth People's Hospital of Shenzhen, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Hebei Provincial Tumor Hospital, Shijiazhuang
  - SuZhou Kowloon Hospital, Suzhou
  - Shanxi Cardiovascular Hospital, Taiyuan
  - The Central Hospital of Tai'an, Tai’an
  - Wu Jing Yi Xue Yuan Fu Shu Yi Yuan, Tianjin
  - Wuhan Asia Heart Hospital, Wuhan
  - Hubei Province Zhongshan Hospital, Wuhan
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Xuzhou Central Hospital, Xuzhou
  - Subei People's Hospital, Yangzhou
  - zhengzhou No.7 people's Hospital, Zhengzhou
  - Zhengzhou Central Hospital, Zhengzhou
  - Zhengzhou People'S Hospital, Zhengzhou
  - Yankuang Group General Hospital, Zoucheng
- Colombia (12):
  - Hospital Santa Clara E.S.E., Bogota DC
  - Fundacion Hospital Infantil Universitario de San José, Bogotá
  - Fundacion Clinica Shaio, Bogotá
  - Simedics Ips, Bogotá
  - Fundacion Valle de Lilly, Cali
  - Centro Médico Julián Coronel, Cali -Valle Del Cauca
  - Centro de Diagnostico Cardilogico, Cartagena
  - Fundacion Cardiovascular de Colombia, Floridablanca
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - Ciclam Sas, Medellín
  - Ces Cardiología, Medellín
  - Fundacion Cardiomet Centro de Investigaciones CEQUIN, Quindío
- Ecuador (3):
  - Hospital Teodoro Maldonado Carbo, Guayaquil
  - Unicormed SA, Guayaquil
  - Hospital INTERVASCU, Quito
- Hong Kong (3):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
- Japan (44):
  - Asahi General Hospital, Chiba, Asahi
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Saiseikai Matsuyama Hospital, Ehime, Matsuyama
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - Japanese Red Cross Fukuoka Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Nakamura Cardiovascular Clinic, Fukuoka, Itoshima
  - Fukuoka Tokushukai Medical Center, Fukuoka, Kasuga
  - Shin Komonji Hospital, Fukuoka, Kitakyushu
  - Fukuoka Shin Mizumaki Hospital, Fukuoka, Onga
  - Matsuda Cardiovascular Clinic, Hokkaido, Sapporo
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Higashi Takarazuka Satoh Hospital, Hyogo, Takarazuka
  - Houju Memorial Hospital, Isikawa, Nomi
  - KKR Takamatsu Hospital, Kagawa , Takamatsu
  - Kagawa Prefectural Shirotori Hospital, Kagawa, Higashikagawa
  - Kokan Clinic, Kanagawa, Kawasaki
  - Sekishinkai Kawasaki Saiwai Clinic, Kanagawa, Kawasaki
  - Sagamihara Kyodo Hospital, Kanagawa, Sagamihara
  - Social Medical Corporation Chikamorikai Chikamori Hospital, Kochi, Kochi
  - Nakayama Clinic of I.M. and Cardiology, Kochi, Cardiology, Kochi, Kochi
  - Sugimurakai Medical Association Sugimura Hospital, Kumamoto, Kumamoto
  - Japan Community Health care Organization Kumamoto General Hospital, Kumamoto, Yatsushiro
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - Iida Municipal Hospital, Nagano, Iida
  - Suwa Red Cross Hospital, Nagano, Suwa
  - Tachikawa General Hospital, Niigata, Nagaoka
  - Nozaki Tokushukai Hospital, Osaka, Daito
  - Teramoto Memorial Hospital, Osaka, Kawachinagano
  - Matsubara Tokushukai Hospital, Osaka, Matsubara
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Kitano Hospital, Osaka, Osaka
  - Osaka Kaisei Hospital, Osaka, Osaka
  - Ishinkai General Clinics, Osaka, Yao
  - Medical corporation Chisei-kai Watanabe clinic, Saitama, Okegawa
  - SAINO Clinic, Saitama, Tokorozawa
  - Kusatsu Heart Center, Shiga, Kusatsu
  - Shizuoka Tokushukai Hospital, Shizuoka, Shizuoka
  - The Institute for Adult Deseases, Asahi Life Foundation, Tokyo, Chuo-ku
  - Minamino Heart Clinic, Tokyo, Hachioji
  - Shimizu Clinic, Tokyo, Kodaira
  - The Cardiovascular Institute Hospital, Tokyo, Minato-ku
  - YOGA Urban Clinic, Tokyo, Setagaya
  - The University of Toyama Hospital, Toyama, Toyama
- Lebanon (10):
  - St.Charles Hospital, Baabda
  - Makassed General Hospital, Beirut
  - St. Georges Hospital, Beirut
  - Hotel Dieu de France Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Al Rassoul Hospital, Beirut Cardiac Institute, Beirut
  - American University of Beirut Medical Center, Beirut
  - Bellvue Medical Center, Beirut, Beirut
  - Notre Dame de Secours Hospital, Byblos
  - Hammoud Hospital University Medical Center, Saida
- Mexico (23):
  - Hospital General de Acapulco, Acapulco de Juárez, Guerrero
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Christius Muguerza Hospital del Parque, Chihuahua City
  - Centro Especializado de Investigación Medical Group Culiacan, Culiacán
  - Centro para el Desarrollo de la Medicina y de Asist Med Espe, Culiacán
  - Instituto Nacional de Cardiologia Ignacio Chavez, Distrito Federal
  - Unidad Coronariana del Hospital General de Durango, Durango
  - Centro de Investigación Especializada de Occidente S.C., Guadalajara
  - Clínica de Estudios Médicos S.C., Guadalajara
  - ICLE SC, Guadalajara
  - Private Practice, Guadalajara
  - Centro Medico de las Americas, Mérida, Yucatán
  - Paracelsus S. A. de C.V., México
  - Hospital Metropolitano "Dr Bernardo Sepulveda", Monterrey
  - Clinica Miravalle, Monterrey, Nuevo Leon
  - Unidad de Investigacion Clinica en Medicina, S.C., Monterrrey
  - Consultorio Privado J Arturo Maldonado Villalon, Morelia, Michoacan
  - Clinical Medical Research S.C, Orizaba
  - Instituto de Corazón de Querétaro, Querétaro
  - Cardioarritmias e Investigación S.C, San Luis Potosí City
  - Plaza Medical, Tijuana
  - Servicios Diagnosticos en Medicina SC, Toluca, Estado de Mexico
  - iBiomed, Zapopan
- Peru (11):
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital Nacional Daniel Alcides Carrion, Bellavista
  - EsSalud - Hospital Nacional IV Alberto Sabogal Sologuren, Callao
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria
  - Hospital Nacional Edgardo Rebaglini Martins, Lima
  - Clinica San Pablo, Lima
  - Centro de Investigación en Diabetes, Obesidad y Nutrición, Lince
  - Clinica Internacional, San Borja
  - Clinica Vesalio, San Borja
  - Clinica El Golf, San Isidro
  - Clinica Medica Cayetano Heredia, San Martín de Porres
- Russia (25):
  - Altaiskyi Reg.Cardiologic Dispensary,Cardiology Dept,Barnaul, Barnaul
  - Chelyabinsk State Med.Acad, Dept. of Clinical Pharmacology, Chelyabinsk
  - Chita State Med.Acad, Consultative-Diagnostic-Polyclinic, Chita
  - OJSC Municipal Instit.Dzerjinskiy City Hospital, Dzerjinskiy
  - Road Clin.Hosp.Irkutsk-Russian Railways,Cardio.&Therapy Dept, Irkutsk
  - City Clin.Hosp.#9,Intern.Diseases&Fam.Practice Dept, Izhevsk, Izhevsk
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - Municipal Instit. City Hosp. No.2, Policlinic Dept,Krasnodar, Krasnodar
  - GOU VPO MUZ City Clinical Hospital No. 20, Krasnoyarsk, Krasnoyarsk
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - Research Center n.a.A.N.Bakulev,Clin.-Diagnostic Dept,Moscow, Moscow
  - Russian Cardiology Research and Production Complex, Moscow, Moscow
  - Reg.Clin.Cardiological Dispen,Arrhythmology Dept,Novosibirsk, Novosibirsk
  - Omsk State Medical Acad.,Internal Diseases&Fam.Practice Dept, Omsk
  - Orenburg State Medical Academy of MoH, Therapy Department, Orenburg
  - Instit.Healthcare,MedicalSanitary Unit 9,n.a.M.A.Tverie,Perm, Perm
  - Rostov Regional Clinical Hospital, Rostov-on-Don
  - Ryazan Reg.Clin.Hosp.Internal Diseases&Policlin.Therapy Dept, Ryazan
  - Fed.Centre of Heart, Blood & Endocrinology n.a. V.A. Almazov, Saint Petersburg
  - Pokrovskaya City Hospital, St.Petersburg, Saint Petersburg
  - Samara Regional Clinical Cardiology Clinic, Day Hosp. Dept., Samara
  - Samara State Medical University, Chair of Faculty Therapy, Samara
  - Municipal Instit.Healthcare,City Policlinic #6,Therapy Dept., Saratov
  - Primorskiy Regional Clinical Hospital No. 1, Vladivostok
  - GBUZ SO Ural Institute of Cardiology, Ekaterinburg, Yekaterinburg
- Saudi Arabia (8):
  - King Fahad Military Hospital, Dammam
  - King Fahad Hufuf Hospital, Hofuf
  - Khamis Military Hospital, Jeddah
  - King Abdul Aziz University Hospital, Jeddah
  - Prince Salman Heart Center, Riyadh
  - King Salman Hospital, Riyadh
  - King Faisal Hospital, Ta'if
  - Tabuk Military Hospital, Tabuk
- Singapore (4):
  - National University Hospital, Singapore
  - National Heart Center, Singapore
  - Novena Heart Centre, Singapore
  - National Neuroscience Institute, Singapore
- South Africa (5):
  - Dr. N. Ranjith, Durban
  - Dr Mahesh Duki Research and Trial Site, Durban
  - LCS Clinical Research Unit, Johannesburg
  - Helderberg Research Institute, Somerset West, Cape Town
  - Dr. Moodley and Dr. Sarvan, Tongaat
- South Korea (31):
  - Sejong General Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National Univ. Hosp, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National Univ. Hosp, Daegu
  - Daegu Fatima Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, Daejeon St.Mary's Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Jeju National University Hospital, Jeju City
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - VHS Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (10):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District
- United Arab Emirates (4):
  - Al Ain Hospital, Abu Dhabi
  - Sheikh Khalifa Medical City, Abu Dhabi
  - Dubai Hospital, Dubai
  - Al Qassimi Hospital, Sharjah city
- Instituto de Clinicas y Urologia Tamanaco, San Roman Caracas, Venezuela

REFERENCES:
- [Derived] Joddrell M, El-Bouri W, Harrison SL, Huisman MV, Lip GYH, Zheng Y; GLORIA-AFinvestigators. Machine learning for outcome prediction in patients with non-valvular atrial fibrillation from the GLORIA-AF registry. Sci Rep. 2024 Nov 7;14(1):27088. doi: 10.1038/s41598-024-78120-z. PMID 39511367
- [Derived] Bergler-Klein J, Gotcheva N, Kalejs O, Kalarus Z, Kovacic D, Persic V, Shlyakhto E, Uuetoa T, Huisman MV, Lip GYH, Vinereanu D; GLORIA-AF Investigators. Antithrombotic Usage, Including Three-Year Outcomes With Dabigatran and Vitamin K Antagonists for Atrial Fibrillation, in Eastern Europe: A Descriptive Analysis From Phase 3 of the GLORIA-AF Registry. Am J Ther. 2024 Jan-Feb 01;31(1):e1-e12. doi: 10.1097/MJT.0000000000001655. Epub 2023 Jan 10. PMID 38231576
- [Derived] Romiti GF, Corica B, Proietti M, Mei DA, Frydenlund J, Bisson A, Boriani G, Olshansky B, Chan YH, Huisman MV, Chao TF, Lip GYH; GLORIA-AF Investigators. Patterns of oral anticoagulant use and outcomes in Asian patients with atrial fibrillation: a post-hoc analysis from the GLORIA-AF Registry. EClinicalMedicine. 2023 Aug 25;63:102039. doi: 10.1016/j.eclinm.2023.102039. eCollection 2023 Sep. PMID 37753446
- [Derived] Ding WY, Fawzy AM, Romiti GF, Proietti M, Pastori D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Validating the predictive ability of the 2MACE score for major adverse cardiovascular events in patients with atrial fibrillation: results from phase II/III of the GLORIA-AF registry. J Thromb Thrombolysis. 2024 Jan;57(1):39-49. doi: 10.1007/s11239-023-02866-y. Epub 2023 Aug 11. PMID 37566295
- [Derived] Liu X, Feng G, Marler SV, Huisman MV, Lip GYH, Ma C. Real world time trends in antithrombotic treatment for newly diagnosed atrial fibrillation in China: reports from the GLORIA-AF Phase III registry : Trends in antithrombotic therapy use in China. Thromb J. 2023 Aug 1;21(1):83. doi: 10.1186/s12959-023-00527-x. PMID 37528405
- [Derived] Ding WY, Lane DA, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Incidence and Risk Factors for Residual Adverse Events Despite Anticoagulation in Atrial Fibrillation: Results From Phase II/III of the GLORIA-AF Registry. J Am Heart Assoc. 2022 Aug 2;11(15):e026410. doi: 10.1161/JAHA.122.026410. Epub 2022 Jul 25. PMID 35876418
- [Derived] Ding WY, Calvert P, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Impact of early ablation of atrial fibrillation on long-term outcomes: results from phase II/III of the GLORIA-AF registry. Clin Res Cardiol. 2022 Sep;111(9):1057-1068. doi: 10.1007/s00392-022-02022-1. Epub 2022 Apr 29. PMID 35488127
- [Derived] Lip GYH, Kotalczyk A, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Marler S, Gurusamy VK, Huisman MV; GLORIA-AF Investigators. Comparative effectiveness and safety of non-vitamin K antagonists for atrial fibrillation in clinical practice: GLORIA-AF Registry. Clin Res Cardiol. 2022 May;111(5):560-573. doi: 10.1007/s00392-022-01996-2. Epub 2022 Mar 16. PMID 35294625
- [Derived] Huisman MV, Teutsch C, Lu S, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Lohmann R, Gurusamy VK, Bartels DB, Lip GYH; GLORIA-AF Investigators. Dabigatran versus vitamin K antagonists for atrial fibrillation in clinical practice: final outcomes from Phase III of the GLORIA-AF registry. Clin Res Cardiol. 2022 May;111(5):548-559. doi: 10.1007/s00392-021-01957-1. Epub 2022 Mar 16. PMID 35294623
- [Derived] Bayer V, Kotalczyk A, Kea B, Teutsch C, Larsen P, Button D, Huisman MV, Lip GYH, Olshansky B. Global Oral Anticoagulation Use Varies by Region in Patients With Recent Diagnosis of Atrial Fibrillation: The GLORIA-AF Phase III Registry. J Am Heart Assoc. 2022 Mar 15;11(6):e023907. doi: 10.1161/JAHA.121.023907. Epub 2022 Mar 4. PMID 35243870
- [Derived] Lopez-Sendon JL, Alonso-Rodriguez D, Baron-Esquivias G, Cosin-Sales J, Marin F, Galera-Llorca J, Jimenez N, Marler S, Huisman MV, Lip GYH; Spanish GLORIA-AF investigators. Gender differences in antithrombotic treatment in patients with atrial fibrillation from Spain versus the rest of Western Europe. GLORIA-AF Program. Med Clin (Barc). 2022 Aug 26;159(4):177-182. doi: 10.1016/j.medcli.2021.09.016. Epub 2021 Dec 8. English, Spanish. PMID 34895750
- [Derived] Ntaios G, Huisman MV, Diener HC, Halperin JL, Teutsch C, Marler S, Gurusamy VK, Thompson M, Lip GYH, Olshansky B; GLORIA-AF Investigators. Anticoagulant selection in relation to the SAMe-TT2R2 score in patients with atrial fibrillation: The GLORIA-AF registry. Hellenic J Cardiol. 2021 Mar-Apr;62(2):152-157. doi: 10.1016/j.hjc.2020.11.009. Epub 2020 Dec 15. PMID 33338644
- [Derived] Mazurek M, Halperin JL, Huisman MV, Diener HC, Dubner SJ, Ma CS, Rothman KJ, Healey JS, Teutsch C, Paquette M, Franca LR, Lu S, Bartels DB, Lip GYH. Antithrombotic treatment for newly diagnosed atrial fibrillation in relation to patient age: the GLORIA-AF registry programme. Europace. 2020 Jan 1;22(1):47-57. doi: 10.1093/europace/euz278. PMID 31651951
- [Derived] Mazurek M, Huisman MV, Rothman KJ, Paquette M, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Zint K, Franca LR, Lu S, Lip GYH; GLORIA-AF Investigators. Gender Differences in Antithrombotic Treatment for Newly Diagnosed Atrial Fibrillation: The GLORIA-AF Registry Program. Am J Med. 2018 Aug;131(8):945-955.e3. doi: 10.1016/j.amjmed.2018.03.024. Epub 2018 Apr 11. PMID 29654720
- [Derived] Huisman MV, Rothman KJ, Paquette M, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Zint K, Elsaesser A, Lu S, Bartels DB, Lip GYH; GLORIA-AF Investigators. Two-year follow-up of patients treated with dabigatran for stroke prevention in atrial fibrillation: Global Registry on Long-Term Antithrombotic Treatment in Patients with Atrial Fibrillation (GLORIA-AF) registry. Am Heart J. 2018 Apr;198:55-63. doi: 10.1016/j.ahj.2017.08.018. Epub 2017 Aug 31. PMID 29653649
- [Derived] Huisman MV, Rothman KJ, Paquette M, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Zint K, Elsaesser A, Bartels DB, Lip GY; GLORIA-AF Investigators. The Changing Landscape for Stroke Prevention in AF: Findings From the GLORIA-AF Registry Phase 2. J Am Coll Cardiol. 2017 Feb 21;69(7):777-785. doi: 10.1016/j.jacc.2016.11.061. PMID 28209218
- [Derived] Huisman MV, Lip GY, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Teutsch C, Zint K, Ackermann D, Clemens A, Bartels DB. Design and rationale of Global Registry on Long-Term Oral Antithrombotic Treatment in Patients with Atrial Fibrillation: a global registry program on long-term oral antithrombotic treatment in patients with atrial fibrillation. Am Heart J. 2014 Mar;167(3):329-34. doi: 10.1016/j.ahj.2013.12.006. Epub 2013 Dec 19. PMID 24576516
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GLORIA-AF was an international, multicentre, non-interventional study based on prospectively collected data for patients (pts) with newly diagnosed non-valvular atrial fibrillation (NVAF). In Ph II, pts baseline characteristics (BC), their antithrombotic treatment patterns and outcomes with 2 years of follow-up for dabigatran alone were collected prospectively. Ph III collected prospective data on pts BC, their treatments and outcomes with 3 years of follow-up for all pts in real-world setting.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the study. Patients attended a participating site which ensured that they (the patients) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Dabigatran Etexilate - Baseline (Phase II): Patients who were prescribed Dabigatran etexilate at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Vitamin K Antagonist (VKA) - Baseline (Phase II): Patients who were prescribed Vitamin K Antagonist (VKA) at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Rivaroxaban - Baseline (Phase II): Patients who were prescribed Rivaroxaban at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Apixaban - Baseline (Phase II): Patients who were prescribed Apixaban at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Acetylsalicylic Acid (ASA) - Baseline (Phase II): Patients who were prescribed Acetylsalicylic acid (ASA) at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Antiplts Other Than ASA - Baseline (Phase II): Patients who were prescribed Antiplts other than Acetylsalicylic acid (ASA) at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- No Treatment - Baseline (Phase II): Patients who were not prescribed any antithrombotic treatments at baseline of Phase II were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Combinations With Oral Anticoagulants - Baseline (Phase II); Combinations With Oral Anticoagulants - Baseline (Phase III): Patients who were prescribed combinations with oral anticoagulants treatments at baseline of Phase III were included in this group. Patients in this group were not included in the safety analysis as no specific treatment can be defined.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Dabigatran Etexilate - Baseline (Phase III): Patients who were prescribed Dabigatran etexilate at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Vitamin K Antagonist (VKA) - Baseline (Phase III): Patients who were prescribed Vitamin K Antagonist (VKA) at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Rivaroxaban - Baseline (Phase III): Patients who were prescribed Rivaroxaban at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Apixaban - Baseline (Phase III): Patients who were prescribed Apixaban at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Edoxaban - Baseline (Phase III): Patients who were prescribed Edoxaban at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Acetylsalicylic Acid (ASA) - Baseline (Phase III): Patients who were prescribed Acetylsalicylic acid (ASA) at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Antiplts Other Than ASA - Baseline (Phase III): Patients who were prescribed Antiplatelets other than ASA at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments may be used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- No Treatment - Baseline (Phase III): Patients who were not prescribed any antithrombotic treatments at baseline of Phase III were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Dabigatran Etexilate - Baseline (Phase II) | Vitamin K Antagonist (VKA) - Baseline (Phase II) | Rivaroxaban - Baseline (Phase II) | Apixaban - Baseline (Phase II) | Acetylsalicylic Acid (ASA) - Baseline (Phase II) | Antiplts Other Than ASA - Baseline (Phase II) | No Treatment - Baseline (Phase II) | Combinations With Oral Anticoagulants - Baseline (Phase II) | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III) | Rivaroxaban - Baseline (Phase III) | Apixaban - Baseline (Phase III) | Edoxaban - Baseline (Phase III) | Acetylsalicylic Acid (ASA) - Baseline (Phase III) | Antiplts Other Than ASA - Baseline (Phase III) | No Treatment - Baseline (Phase III) | Combinations With Oral Anticoagulants - Baseline (Phase III)
Started | 4964 | 5103 | 1784 | 715 | 1736 | 128 | 1209 | 5 | 3879 | 4962 | 4054 | 4538 | 333 | 2182 | 214 | 1418 | 11
All Eligible Patient | 4873 | 4963 | 1755 | 703 | 1714 | 126 | 1170 | 4 | 3839 | 4836 | 4015 | 4505 | 332 | 2163 | 213 | 1386 | 11
Completed | 3965 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3219 | 3780 | 3256 | 3672 | 284 | 1712 | 151 | 1056 | 10
Not Completed | 999 | 5103 | 1784 | 715 | 1736 | 128 | 1209 | 5 | 660 | 1182 | 798 | 866 | 49 | 470 | 63 | 362 | 1
Not completed — Not eligible | 91 | 140 | 29 | 12 | 22 | 2 | 39 | 1 | 40 | 126 | 39 | 33 | 1 | 19 | 1 | 32 | 0
Not completed — Lost to Follow-up | 306 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 215 | 309 | 224 | 212 | 11 | 164 | 17 | 127 | 1
Not completed — Withdrawal by Subject | 165 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 83 | 88 | 100 | 114 | 9 | 47 | 6 | 31 | 0
Not completed — Other reasons than listed | 437 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 318 | 658 | 433 | 504 | 28 | 239 | 39 | 172 | 0
Not completed — No end of study case report form | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Not being followed up | 0 | 4963 | 1755 | 703 | 1714 | 126 | 1170 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible: All patients who were enrolled and eligible (i.e. did not have any important. protocol violation(s) and who met certain data cleaning requirements).
Groups:
- Combinations With Oral Anticoagulants - Baseline (Phase II): Patients who were prescribed combinations with oral anticoagulants treatments at baseline of Phase II were included in this group. Patients in this group were not included in the safety analysis as no specific treatment can be defined.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate - Baseline (Phase II) | Vitamin K Antagonist (VKA) - Baseline (Phase II) | Rivaroxaban - Baseline (Phase II) | Apixaban - Baseline (Phase II) | Acetylsalicylic Acid (ASA) - Baseline (Phase II) | Antiplts Other Than ASA - Baseline (Phase II) | No Treatment - Baseline (Phase II) | Combinations With Oral Anticoagulants - Baseline (Phase II) | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III) | Rivaroxaban - Baseline (Phase III) | Apixaban - Baseline (Phase III) | Edoxaban - Baseline (Phase III) | Acetylsalicylic Acid (ASA) - Baseline (Phase III) | Antiplts Other Than ASA - Baseline (Phase III) | No Treatment - Baseline (Phase III) | Combinations With Oral Anticoagulants - Baseline (Phase III) | Total
Number analyzed (Participants) | 4873 | 4963 | 1755 | 703 | 1714 | 126 | 1170 | 4 | 3839 | 4836 | 4015 | 4505 | 332 | 2163 | 213 | 1386 | 11 | 36608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (10.4) | 71.4 (10.6) | 71.5 (10.6) | 73.8 (10.0) | 67.7 (12.4) | 73.5 (10.7) | 68.3 (12.5) | 76.0 (8.3) | 70.1 (10.2) | 71.2 (10.3) | 70.3 (10.2) | 72.4 (10.1) | 72.3 (9.4) | 68.0 (11.8) | 73.1 (10.8) | 67.6 (12.2) | 70.2 (12.1) | 70.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2162 | 2304 | 773 | 338 | 778 | 58 | 553 | 2 | 1718 | 2152 | 1766 | 2104 | 139 | 931 | 92 | 660 | 6 | 16536
  Male | 2711 | 2659 | 982 | 365 | 936 | 68 | 617 | 2 | 2121 | 2684 | 2249 | 2401 | 193 | 1232 | 121 | 726 | 5 | 20072
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 14 | 6 | 0 | 4 | 0 | 1 | 0 | 27 | 32 | 32 | 21 | 0 | 7 | 2 | 3 | 1 | 170
  Asian | 423 | 797 | 111 | 93 | 694 | 43 | 603 | 0 | 841 | 760 | 381 | 413 | 125 | 916 | 95 | 593 | 8 | 6896
  Black/African American | 40 | 86 | 42 | 14 | 44 | 0 | 23 | 0 | 47 | 85 | 72 | 118 | 2 | 49 | 2 | 23 | 0 | 647
  Native Hawaiian/Other Pacific Islander | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 9
  White | 3372 | 3590 | 1375 | 538 | 863 | 70 | 497 | 4 | 2484 | 3611 | 3126 | 3528 | 203 | 1057 | 104 | 708 | 2 | 25132
  Other | 447 | 262 | 69 | 24 | 82 | 10 | 21 | 0 | 181 | 144 | 144 | 79 | 2 | 57 | 7 | 32 | 0 | 1561
  Missing | 571 | 211 | 151 | 34 | 26 | 3 | 24 | 0 | 259 | 204 | 260 | 345 | 0 | 75 | 3 | 27 | 0 | 2193

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction, Life-threatening Bleeding Events and Vascular Death) - Phase II
Description: Incidence rate of composite outcome which includes events of Stroke, systemic embolism, myocardial infarction, life-threatening bleeding events and vascular death on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only. In case of multiple events for a patient, the first event was considered.
Time Frame: From baseline visit of Phase II until end of initial treatment regimen episode (minimum date of permanent stop of DE + 3 days, start date of other treatments - 1 day, and date of study completion/discontinuation), up to 2 years.
Population: All eligible patients who were prescribed DE at baseline in phase II excluding prescribed but not taken. All eligible: All patients who were enrolled and eligible (i.e. did not have any important. protocol violation(s) and who met certain data cleaning requirements).
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 2.06 [1.74 to 2.42]

2. Primary Outcome: Incidence Rate of Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction, Life-threatening Bleeding Events and Vascular Death) - Phase III
Description: Incidence rate of composite outcome which includes events of Stroke, systemic embolism, myocardial infarction, life-threatening bleeding events and vascular death on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only. In case of multiple events for a patient, the first event was considered. Unknown cause of death was imputed by multiple imputation. Counts were based on the average of the 20 restricted data sets. The average of the 20 incidence rates from the 20 imputed datasets were used to obtain the point estimate of the incidence rate that is reported here. The bootstrapping approach was used to obtain the 95% confidence interval of the incidence rate.
Time Frame: From baseline visit of phase III until end of initial treatment regimen episode (minimum date of permanent stop of DE + 3 days/ VKA+ 6 days, start date of other treatments - 1 day, and date of study completion/discontinuation), up to 3 years.
Population: Restricted patient set: was defined only for eligible dabigatran and vitamin K antagonist patients (pts) of phase III who were within region of propensity score (PS) overlap excluding pts in non-overlapping tails of PS distribution, using cut-offs at 1.5th percentile of the PS distribution for dab-exposed group, and 98.5th percentile of distribution for VKA-exposed group. Excluding these pts from the tails of PS distribution reduces channeling bias and improves the validity of comparisons.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Groups:
- Vitamin K Antagonist (VKA) - Baseline (Phase III): Patients who were prescribed at baseline of Phase III the Vitamin K Antagonist (VKA) were included in this group. Patients could take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments may used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 2.21 [1.88 to 2.57] | 3.23 [2.83 to 3.62]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous stroke/transient ischaemic attack/systemic embolism, previous myocardial infarction, abnormal kidney function and concomitant antiplatelets use; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.90] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

3. Primary Outcome: Incidence Rate of Vascular Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction and Vascular Death) - Phase II
Description: Incidence rate of vascular composite outcome including events of stroke, systemic embolism, myocardial infarction and vascular death on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only. In case of multiple events for a patient, the first event was considered.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 1.74 [1.45 to 2.07]

4. Primary Outcome: Incidence Rate of Vascular Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction and Vascular Death) - Phase III
Description: Incidence rate of vascular composite outcome including events of stroke, systemic embolism, myocardial infarction and vascular death on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only. In case of multiple events for a patient, the first event was considered. Unknown death was imputed by multiple imputation. Counts were based on the average of the 20 restricted data sets. The average of the 20 incidence rates from the 20 imputed datasets were used to obtain the point estimate of the incidence rate that is reported here. The bootstrapping approach was used to obtain the 95% confidence interval of the incidence rate.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 1.91 [1.59 to 2.24] | 2.62 [2.27 to 2.96]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); [analysis description as in outcome 2, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.63 to 0.98] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

5. Primary Outcome: Incidence Rate of Stroke or Systemic Embolism - Phase III
Description: Incidence rate of stroke or systemic embolism on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.80 [0.61 to 1.01] | 1.00 [0.80 to 1.22]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); [analysis description as in outcome 2, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.11] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

6. Primary Outcome: Incidence Rate of Stroke - Phase II
Description: Incidence rate of stroke on all eligible patients excluding prescribed but not taken set for Dabigatran etexilate (DE) of phase II only is presented. Stroke is an acute onset of a focal neurological deficit of presumed vascular origin lasting for 24 hours or more or resulting in death. The stroke included ischemic or hemorrhagic or uncertain classification.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.65 [0.48 to 0.87]

7. Primary Outcome: Incidence Rate of Stroke - Phase III
Description: Incidence rate of stroke on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only. Stroke is an acute onset of a focal neurological deficit of presumed vascular origin lasting for 24 hours or more or resulting in death. The stroke included ischemic or hemorrhagic or uncertain classification.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.77 [0.58 to 0.97] | 0.96 [0.76 to 1.17]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); [analysis description as in outcome 2, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.57 to 1.14] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

8. Primary Outcome: Incidence Rate of Transient Ischaemic Attack (TIA) - Phase II
Description: Incidence rate of transient ischaemic attack (TIA) on on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.21 [0.12 to 0.34]

9. Primary Outcome: Incidence Rate of Transient Ischaemic Attack (TIA) - Phase III
Description: Incidence rate of transient ischaemic attack (TIA) on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.29 [0.17 to 0.42] | 0.32 [0.21 to 0.45]

10. Primary Outcome: Incidence Rate of Systemic Embolism (SE) - Phase II
Description: Incidence rate of systemic embolism (SE) on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.04 [0.01 to 0.12]

11. Primary Outcome: Incidence Rate of Systemic Embolism (SE) - Phase III
Description: Incidence rate of systemic embolism (SE) on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.04 [0.00 to 0.09] | 0.05 [0.01 to 0.09]

12. Primary Outcome: Incidence Rate of Pulmonary Embolism (PE) - Phase II
Description: Incidence rate of pulmonary embolism (PE) on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.07 [0.02 to 0.16]

13. Primary Outcome: Incidence Rate of Pulmonary Embolism (PE) - Phase III
Description: Incidence rate of pulmonary embolism (PE) on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.07 [0.01 to 0.13] | 0.06 [0.01 to 0.11]

14. Primary Outcome: Incidence Rate of Major Bleeding Events (MBE) - Phase II
Description: Incidence rate of major bleeding events (MBE) on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented. Major bleeding was defined as meeting one or more of the following criteria: Overt bleeding associated with a reduction in haemoglobin of at least 20 grams per liter or leading to a transfusion of at least 2 units of blood or packed cells; Symptomatic bleeding in a critical area or organ: Intraocular, intracranial, intraspinal or intramuscular with compartment syndrome, retroperitoneal bleeding, intra-articular bleeding or pericardial bleeding; Life-threatening bleeding.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.97 [0.76 to 1.23]

15. Primary Outcome: Incidence Rate of Major Bleeding Events (MBE) - Phase III
Description: Incidence rate of major bleeding events on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only. Major bleeding was defined as meeting one or more of the following criteria: Overt bleeding associated with a reduction in haemoglobin of at least 20 grams per liter or leading to a transfusion of at least 2 units of blood or packed cells; Symptomatic bleeding in a critical area or organ: Intraocular, intracranial, intraspinal or intramuscular with compartment syndrome, retroperitoneal bleeding, intra-articular bleeding or pericardial bleeding; Life-threatening bleeding.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.69 [0.51 to 0.89] | 1.44 [1.20 to 1.70]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous myocardial infarction, abnormal kidney function, concomitant antiplatelets use and concomitant use of drugs related to bleeding; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.38 to 0.73] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

16. Primary Outcome: Incidence Rate of Life-threatening Bleeding Events - Phase II
Description: Incidence rate of life-threatening bleeding events on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented. Life-threatening bleeding was defined as meeting one or more of the following criteria: Symptomatic intracranial bleed; Reduction in haemoglobin of at least 50 grams per liter; Transfusion of at least 4 units of blood or packed cells, associated with hypotension requiring the use of intravenous inotropic agents; Necessitated surgical intervention; Fatal bleeding.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.46 [0.32 to 0.64]

17. Primary Outcome: Incidence Rate of Life-threatening Bleeding Events - Phase III
Description: Incidence rate of life-threatening bleeding events on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only. Life-threatening bleeding was defined as meeting one or more of the following criteria: Symptomatic intracranial bleed; Reduction in haemoglobin of at least 50 grams per liter; Transfusion of at least 4 units of blood or packed cells, associated with hypotension requiring the use of intravenous inotropic agents; Necessitated surgical intervention; Fatal bleeding.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.47 [0.32 to 0.63] | 1.07 [0.86 to 1.30]

18. Primary Outcome: Incidence Rate of Myocardial Infarction (MI) - Phase II
Description: Incidence rate of myocardial infarction (MI) on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.50 [0.35 to 0.69]

19. Primary Outcome: Incidence Rate of Myocardial Infarction (MI) - Phase III
Description: Incidence rate of myocardial infarction on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.40 [0.27 to 0.55] | 0.53 [0.38 to 0.68]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous myocardial infarction, concomitant antiplatelets use, concomitant use of drugs related to bleeding, hypertension, and diabetes; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.60 to 1.57] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

20. Primary Outcome: Incidence Rate of All-cause Death - Phase II
Description: Incidence rate of all-cause death on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 2.48 [2.13 to 2.87]

21. Primary Outcome: Incidence Rate of All-cause Death - Phase III
Description: Incidence rate of all-cause death on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 2.16 [1.84 to 2.48] | 3.57 [3.19 to 3.96]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline (Phase III) vs Vitamin K Antagonist (VKA) - Baseline (Phase III); [analysis description as in outcome 2, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.54 to 0.80] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

22. Primary Outcome: Incidence Rate of Vascular Death - Phase II
Description: Incidence rate of vascular death on all eligible patients excluding prescribed but not taken set that included Dabigatran etexilate (DE) of phase II only is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase II)
Number analyzed (Participants) | 4859
Events per 100 person-years | 0.85 [0.65 to 1.09]

23. Primary Outcome: Incidence Rate of Vascular Death - Phase III
Description: Incidence rate of vascular death on restricted set that included Dabigatran etexilate (DE) of phase III and Vitamin K Antagonist (VKA) of phase III only.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline (Phase III) | Vitamin K Antagonist (VKA) - Baseline (Phase III)
Number analyzed (Participants) | 3611 | 4413
Events per 100 person-years | 0.75 [0.56 to 0.95] | 1.26 [1.03 to 1.50]

ADVERSE EVENTS:
Time Frame: Phase (Ph) II: From baseline visit of Phase II until Phase II completion or discontinuation, up to 2 years of follow-up. Only patients who were prescribed Dabigatran etexilate at baseline of Phase II were followed up. Phase III: From baseline visit of Phase III until study completion or discontinuation, up to 3 years of follow-up for all patients irrespective of their antithrombotic treament.
Description: Enrolled+treated: Patients(pts) entered electronic data system who signed informed consent+treated at least once with study treatments(trt). Only trt-related AEs collected +reported according to protocol-specified requirements. PhII: only AEs for pts who presribed DE at baseline collected+reported. PhIII:"Combinations of oral anticoagulants at baseline" excluded as no specific trt could be defined for AEs that occurred on trt interval on which they were on combination of oral anticoagulants.
Groups:
- Dabigatran Etexilate - at Least Once During Phase III of the Study: All patients who received at least once dabigatran etexilate during phase III of the study were included in the group. Adverse events which happened when the patients received dabigatran etexilate were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Vitamin K Antagonist (VKA) - at Least Once During Phase III of the Study: All patients who received at least once Vitamin K Antagonist (VKA) during phase III of the study were included in the group. Adverse events which happened when the patients received Vitamin K Antagonist (VKA) were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Rivaroxaban - at Least Once During Phase III of the Study: All patients who received at least once Rivaroxaban during phase III of the study were included in the group. Adverse events which happened when the patients received Rivaroxaban were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Apixaban - at Least Once During Phase III of the Study: All patients who received at least once Apixaban during phase III of the study were included in the group. Adverse events which happened when the patients received Apixaban were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Edoxaban - at Least Once During Phase III of the Study: All patients who received at least once Edoxaban during phase III of the study were included in the group. Adverse events which happened when the patients received Edoxaban were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Acetylsalicylic Acid (ASA) - at Least Once During Phase III of the Study: All patients who received at least once Acetylsalicylic acid (ASA) during phase III of the study were included in the group. Adverse events which happened when the patients received Acetylsalicylic acid (ASA) were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Antiplts Other Than ASA - at Least Once During Phase III of the Study: All patients who received at least once Antiplts other than ASA during phase III of the study were included in the group. Adverse events which happened when the patients received Antiplts other than ASA were reported in this group.
  Patients can take any Antithrombotic treatments during phase III of the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
Arm/Group | Dabigatran Etexilate - Baseline (Phase II) | Dabigatran Etexilate - at Least Once During Phase III of the Study | Vitamin K Antagonist (VKA) - at Least Once During Phase III of the Study | Rivaroxaban - at Least Once During Phase III of the Study | Apixaban - at Least Once During Phase III of the Study | Edoxaban - at Least Once During Phase III of the Study | Acetylsalicylic Acid (ASA) - at Least Once During Phase III of the Study | Antiplts Other Than ASA - at Least Once During Phase III of the Study
All-Cause Mortality (participants affected / at risk) | 184/4943 | 199/4477 | 465/5894 | 292/5177 | 392/6024 | 23/686 | 469/6263 | 46/780
Serious Adverse Events (participants affected / at risk) | 985/4943 | 118/4477 | 296/5894 | 185/5177 | 217/6024 | 16/686 | 225/6263 | 19/780
Other Adverse Events (participants affected / at risk) | 0/4943 | 0/4477 | 0/5894 | 0/5177 | 0/6024 | 0/686 | 0/6263 | 0/780
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dabigatran Etexilate - Baseline (Phase II) (N=4943) | Dabigatran Etexilate - at Least Once During Phase III of the Study (N=4477) | Vitamin K Antagonist (VKA) - at Least Once During Phase III of the Study (N=5894) | Rivaroxaban - at Least Once During Phase III of the Study (N=5177) | Apixaban - at Least Once During Phase III of the Study (N=6024) | Edoxaban - at Least Once During Phase III of the Study (N=686) | Acetylsalicylic Acid (ASA) - at Least Once During Phase III of the Study (N=6263) | Antiplts Other Than ASA - at Least Once During Phase III of the Study (N=780)
Anaemia (Blood and lymphatic system disorders) | 12 | 6 | 16 | 12 | 19 | 2/636 | 19 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 2 | 9 | 4 | 4 | 1/636 | 7 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0/636 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3 | 1 | 0/636 | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0/636 | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0/636 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 0/636 | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Angina pectoris (Cardiac disorders) | 20 | 1 | 1 | 0 | 0 | 0/636 | 1 | 0
Angina unstable (Cardiac disorders) | 11 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 159 | 0 | 3 | 2 | 1 | 0/636 | 3 | 0
Atrial flutter (Cardiac disorders) | 9 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 3 | 0 | 1 | 1 | 0 | 0/636 | 0 | 0
Bradycardia (Cardiac disorders) | 14 | 0 | 2 | 0 | 0 | 0/636 | 1 | 0
Cardiac arrest (Cardiac disorders) | 9 | 1 | 0 | 1 | 1 | 0/636 | 1 | 0
Cardiac failure (Cardiac disorders) | 67 | 3 | 4 | 0 | 2 | 0/636 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 41 | 1 | 1 | 0 | 0 | 0/636 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1 | 0 | 0 | 2 | 0/636 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Cardiomyopathy alcoholic (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Myocardial infarction (Cardiac disorders) | 27 | 2 | 2 | 1 | 0 | 0/636 | 2 | 0
Palpitations (Cardiac disorders) | 9 | 0 | 1 | 1 | 0 | 0/636 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Pericardial haemorrhage (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0/636 | 1 | 0
Pericarditis (Cardiac disorders) | 4 | 0 | 0 | 1 | 0 | 0/636 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 0 | 0 | 1 | 0 | 0/636 | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 1 | 0 | 2 | 0/636 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Retinal vascular occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0/636 | 2 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 0/636 | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0/636 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0/636 | 2 | 0
Discoloured vomit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 1 | 1/636 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0/636 | 2 | 0
Duodenal varices (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2 | 0/636 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3 | 0/636 | 3 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 3 | 1/636 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 24 | 16 | 27 | 36 | 26 | 3/636 | 43 | 4
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 1 | 0/636 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 3 | 0 | 2 | 3 | 0/636 | 4 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 1 | 0/636 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0/636 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0/636 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 12 | 11 | 21 | 10 | 1/636 | 20 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 2 | 0/636 | 2 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 2 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0/636 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 8 | 6 | 8 | 6 | 7 | 2/636 | 8 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0/636 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 8 | 18 | 8 | 12 | 0/636 | 9 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Vomiting projectile (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0/636 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 2 | 0 | 0/636 | 1 | 2
Medical device site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 0/636 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0/636 | 2 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 1 | 0/636 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0/636 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cellulitis (Infections and infestations) | 7 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0/636 | 1 | 0
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0/636 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0/636 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Pneumonia (Infections and infestations) | 41 | 1 | 0 | 2 | 2 | 0/636 | 0 | 0
Sepsis (Infections and infestations) | 9 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 1 | 1 | 0 | 0 | 0/636 | 1 | 0
Urosepsis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0/636 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0/636 | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 1 | 8 | 2 | 4 | 0/636 | 5 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 6 | 0 | 1 | 0/636 | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2 | 0/636 | 2 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0/636 | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 5 | 1 | 0/636 | 4 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 0/636 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0/636 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 0/636 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 4 | 13 | 0 | 2 | 0/636 | 7 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 1 | 1 | 0/636 | 2 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 9 | 0 | 0 | 0/636 | 4 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0/636 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1/636 | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0/636 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 7 | 0 | 0 | 0/636 | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Blood urine present (Investigations) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Catheterisation cardiac (Investigations) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0/636 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 7 | 1 | 1 | 0/636 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Occult blood (Investigations) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0/636 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 0/636 | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 0 | 1 | 0/636 | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 4 | 0/636 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0/636 | 1 | 0
Sarcomatoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0/636 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1/636 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 1 | 10 | 3 | 5 | 1/636 | 5 | 0
Cerebral infarction (Nervous system disorders) | 7 | 1 | 1 | 1 | 2 | 0/636 | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 20 | 0 | 9 | 1 | 7 | 0/636 | 5 | 0
Dizziness (Nervous system disorders) | 7 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2/636 | 3 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 1 | 10 | 4 | 2 | 0/636 | 5 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 2 | 7 | 4 | 5 | 0/636 | 2 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0/636 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 19 | 7 | 9 | 3 | 5 | 0/636 | 6 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 1 | 0
Presyncope (Nervous system disorders) | 3 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1 | 3 | 2 | 4 | 0/636 | 2 | 0
Syncope (Nervous system disorders) | 18 | 0 | 1 | 2 | 1 | 0/636 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 15 | 5 | 13 | 5 | 7 | 0/636 | 5 | 0
Vascular dementia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0 | 0 | 1 | 1 | 0/636 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 3 | 12 | 10 | 5 | 0/636 | 6 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0/636 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1 | 7 | 1 | 2 | 0/636 | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1/636 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 0 | 3 | 1 | 0/636 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 1 | 0 | 0 | 4 | 0/636 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 19 | 8 | 8 | 1/636 | 8 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 5 | 1 | 5 | 0/636 | 4 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0/636 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0/636 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2 | 0 | 0 | 0/636 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0/636 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 10 | 1 | 4 | 0/636 | 3 | 1
Haemorrhage (Vascular disorders) | 0 | 3 | 8 | 4 | 10 | 0/636 | 4 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 2 | 0 | 0 | 0/636 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0/636 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0/636 | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0/636 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 0/636 | 0 | 0
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Venous haemorrhage (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0/636 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/636 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0/636 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Normochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 8 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Arrhythmia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 5 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiac disorder (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 5 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Coronary artery disease (Cardiac disorders) | 7 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Left ventricular failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Myocardial fibrosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sinoatrial block (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sinus arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 16 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 5 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 5 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Thyroid mass (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tooth pulp haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cardiac death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Death (General disorders) | 48 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gait disturbance (General disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Non-cardiac chest pain (General disorders) | 10 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Organ failure (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sudden death (General disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ulcer (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Arthritis infective (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Echinococciasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Endocarditis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Erysipelas (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Paraspinal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Septic arthritis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Septic shock (Infections and infestations) | 7 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Viral infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pocket erosion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Procedural shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Malignant genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dementia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dysarthria (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Epilepsy (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Intracranial mass (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Spinal cord haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Device battery issue (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Device dislocation (Product Issues) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Device loosening (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Device malfunction (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Derailment (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Renal aneurysm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Renal failure (Renal and urinary disorders) | 12 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Renal impairment (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Alcoholic (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Aortic stenosis (Vascular disorders) | 6 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypertension (Vascular disorders) | 11 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0/636 | 0 | 0

LIMITATIONS AND CAVEATS:
Phase II part of 1160.129 includes Phase II data from 1160.129, 1160.136 and 1160.171.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT01468701/SAP_000.pdf
  • Study Protocol (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT01468701/Prot_001.pdf